CLINICAL TRIAL: NCT02755818
Title: The Independent Effect of Level of Kidney Function and Body Composition On Establishing HDL Cholesterol Levels
Brief Title: Study of the Relationship Between Body Composition, Insulin Resistance and HDL Levels
Status: Terminated | Type: Observational
Why Stopped: insufficient patients with CKD willing to be injected with heparin
Sponsor: University of California, Davis (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 220939
Record Dates: First submitted 2016-03-10; First posted 2016-04-29 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: high density lipoprotein (HDL); lipid; insulin resistance; glomerular filtration rate (GFR); obesity
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood taken separated into plasma, serum, and red cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control: heparin at 50unit/kg of body weight having glomerular filtration rate (GFR) of greater than 60
  Interventions: Drug: Heparin
- chronic renal disease (CKD3b): heparin at 50unit/kg of body weight having glomerular filtration rate (GFR) of 30-45
  Interventions: Drug: Heparin
- chronic renal disease (CKD4): heparin at 50unit/kg of body weight having glomerular filtration rate (GFR) of 15-30
  Interventions: Drug: Heparin
- chronic renal disease (CKD5): heparin at 50unit/kg of body weight having glomerular filtration rate (GFR) of less than 15, or on hemodialysis
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin — This is not an interventional study. The investigators use heparin at 50unit/kg of body weight to release enzyme lipoprotein lipase (LPL) from the body. LPL level will be used as part of calculation of lipid analysis and measurements
  Other Names: Heparin Sodium

SUMMARY:
Approximately 20 million people in the United States have some form of kidney failure. People with kidney failure have an increased chance of having low levels of high density lipid (HDL), so called "good cholesterol." Patients who are overweight or obese also have low levels of HDL. The investigators are trying to find out whether causes of low HDL are the same in people who are overweight and in patients with kidney failure so that in the future doctors can better treat low HDL cholesterol levels. People with low levels of HDL are more likely to have heart attacks and strokes and are more likely to lose kidney function. This study hope to learn more about how kidney failure causes low HDL cholesterol levels.

DETAILED DESCRIPTION:
This study is not a treatment or outcome trial.This is a single center cross sectional analysis of body composition and lipoprotein level and structure among patients with graded levels of renal failure in comparison to control subjects. To study the relationship between HDL cholesterol and both body composition and insulin resistance measured as homeostatic model assessment (HOMA) among a cohort of non diabetic non-proteinuric patients with advanced chronic kidney disease (CKD) compared to non diabetic subjects having normal kidney function. Renal patients chosen will be with advanced CKD stage 3, Stage 4, and stage 5 - which is end stage renal failure (ESRD) and on hemodialysis. Fasting blood will be taken for the evaluation of baseline lipid and renal function, and blood glucose level to make sure that there is no recent evidence of diabetes. Body compositions will be measured with 2 established methods: DEXA and whole body bio-impedance spectroscopy (BIS). Fat mass and analysis will be estimated so as to provide a relationship between adiposity, insulin resistance, residual renal function and HDL levels and structure.

ELIGIBILITY:
Inclusion Criteria:

* self report of stable body weight during the past six months;
* BMI 18-40 kg/m2; Hemodialysis dependent for at least 3 months, prevalent ESRD (end stage renal disease) cohort;
* GFR > 15 < 44 ml/min (CKD cohort);
* GFR > 60 ml/min (Control cohort).

Exclusion Criteria:

* Diabetes Mellitus (American Diabetes Association definition: fasting glucose >120 mg/dl);
* Evidence of liver disorder, ie; hepatitis
* Evidence of thyroid disorders
* HIV by medical history (HIV test will not be performed)
* Renal transplant recipient
* Oral contraceptive/ hormone replacement therapy
* Systemic use of systemic or inhaled corticosteroids in the past month
* Contraindication to systemic anticoagulation (heparin administration is necessary to measure levels of LPL, HL);
* Hemoglobin < 8.5 g/dl (anemia);
* Current, within 2 months use of any hypolipidemic or anti-diabetic agents;
* Patients treated with a fibric acid derivative or niacin in the past 4 weeks;
* Urinary protein excretion of greater than 0.5 grams per day;
* Any other condition that, in the opinion of the investigators, would put the subject at risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a single center cross sectional study of renal failure in comparison to control subjects. This is not a treatment or outcome trial.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-10-22 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Kaysen, MD PhD, Principal Investigator — University of California, Davis; Tjien Dwyer, BS, Study Director — University of California, Davis

IPD SHARING:
Plan to Share IPD: Yes
once published; data will be shared
Supporting Information: SAP, ICF
Time Frame: once published; data will be shared
Access Criteria: once published; data will be shared

REFERENCES:
- [Result] Molfino A, Don BR, Kaysen GA. Comparison of bioimpedance and dual-energy x-ray absorptiometry for measurement of fat mass in hemodialysis patients. Nephron Clin Pract. 2012;122(3-4):127-33. doi: 10.1159/000350817. Epub 2013 May 9. PMID 23689544
- See also: Nephron Clin Pract. 2012; 122(0): 127-133. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4353643/
- Available data/document: Informed Consent Form — https://www.irbnet.org/release/study/overview.do?ctx_id=0&spk_id=855867 — for a copy of Approved Consent Form-please contact Study Coordinator -Tjien Dwyer at tlthio@ucdavis.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects are recruited from Sacramento areas within 50 miles radius, and University of California, Davis. Subjects of chronic kidney disease (CKD5) are recruited mainly from five DCI (Dialysis Clinic Incorporation) clinics in Sacramento area.
Period: Overall Study
Arm/Group | Control | Chronic Renal Disease (CKD3b) | Chronic Renal Disease (CKD4) | Chronic Renal Disease (CKD5)
Started | 30 | 2 | 2 | 17
Completed | 30 | 2 | 1 | 14
Not Completed | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — withdrawal by PI | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Non-diabetic
Groups:
- Chronic Renal Disease (CKD3b): heparin at 50unit/kg of body weight having glomerular filtration rate (GFR) of greater than 30-45
  Heparin: This is not an interventional study. The investigators use heparin at 50unit/kg of body weight to release enzyme lipoprotein lipase (LPL) from the body. LPL level will be used as part of calculation of lipid analysis and measurements
- Chronic Renal Disease (CKD4): heparin at 50unit/kg of body weight having glomerular filtration rate (GFR) of greater than 15-30
  Heparin: This is not an interventional study. The investigators use heparin at 50unit/kg of body weight to release enzyme lipoprotein lipase (LPL) from the body. LPL level will be used as part of calculation of lipid analysis and measurements
- Total: Total of all reporting groups
Arm/Group | Control | Chronic Renal Disease (CKD3b) | Chronic Renal Disease (CKD4) | Chronic Renal Disease (CKD5) | Total
Number analyzed (Participants) | 30 | 2 | 2 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 0 | 2 | 17 | 49
  >=65 years | 0 | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 0 | 2 | 3 | 21
  Male | 14 | 2 | 0 | 14 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 1 | 0 | 0 | 6
  African American | 3 | 0 | 1 | 8 | 12
  Hispanic | 6 | 0 | 0 | 3 | 9
  Non-Hispanic | 15 | 1 | 1 | 6 | 23
  Other | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: HDL (High Density Lipoprotein) Level in Control and Chronic Kidney Disease (CKD 3b, 4, 5) Groups
Description: HDL (high-density lipoprotein), is called "good" cholesterol. It binds to cholesterols marked for disposal back to the liver to be digested and disposed by the body. High HDL level may lower your risk for heart disease and stroke.
Time Frame: HDL (high density lipoprotein) (mg/dL) -- this is a cross sectional study; only one measurement collected, termed "baseline"
Population: Data missing (1) for CKD4 group
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Control: Subject has glomerular filtration rate (GFR) of greater than 60 cc/min -- indication of normal kidney
- Chronic Kidney Disease, Stage 5 (CKD5): Subject has glomerular filtration rate (GFR) of less than 15 cc/min - all subjects are on kidney dialysis
- Chronic Kidney Disease 4 (CKD4): Subject has glomerular filtration rate (GFR) of 15-29 cc/min
- Chronic Kidney Disease Stage 3b (CKD 3b): Subject has glomerular filtration rate (GFR) of 30-45 cc/min
Arm/Group | Control | Chronic Kidney Disease, Stage 5 (CKD5) | Chronic Kidney Disease 4 (CKD4) | Chronic Kidney Disease Stage 3b (CKD 3b)
Number analyzed (Participants) | 30 | 14 | 1 | 2
mg/dL | 46.77 (14.88) | 38.79 (11.9) | 71 (NA) — only 1 participant - standard deviation not calculated | 43.50 (9.19)

2. Primary Outcome: LDL Level in Control and Chronic Kidney Disease (CKD3b, CKD4, CKD5) Groups
Description: LDL (low-density lipoprotein), is a type of cholesterol (fat) circulating in the blood vessels, and can form plaques. High levels of LDL cholesterol may raise your risk for heart disease and stroke.
Time Frame: This is a cross sectional study; only one measurement collected, termed "baseline"
Population: Data missing (1) for CKD4 group
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Chronic Kidney Disease, Stage 4 (CKD4): Subject has glomerular filtration rate (GFR) of 15-29 cc/min - subject has severe kidney disease
- Chronic Kidney Disease, Stage 3b (CKD3b): Subject has glomerular filtration rate (GFR) of 30-44 cc/min - subject has markedly reduced kidney function
Arm/Group | Control | Chronic Kidney Disease, Stage 5 (CKD5) | Chronic Kidney Disease, Stage 4 (CKD4) | Chronic Kidney Disease, Stage 3b (CKD3b)
Number analyzed (Participants) | 30 | 14 | 1 | 2
mg/dL | 105.93 (28.03) | 75.29 (25.17) | 235 (NA) — one patient only- no standard deviation calculated | 112.50 (30.41)

3. Primary Outcome: C Reactive Protein (CRP) Level in Control and Chronic Kidney Disease (CKD3b, CKD4, CKD5) Groups
Description: C-reactive protein (CRP) is an inflammation marker produced by the liver. An increase in CRP value may means inflammation in the body.
Time Frame: This is a cross sectional study; only one measurement collected, termed "baseline"
Population: Data missing (1) for CKD4 group
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Chronic Kidney Disease, Stage 5 (CKD5) | Chronic Kidney Disease, Stage 4 (CKD4) | Chronic Kidney Disease, Stage 3b (CKD3b)
Number analyzed (Participants) | 30 | 14 | 1 | 2
mg/dL | 0.26 (0.17) | 0.74 (0.64) | 1.6 (NA) — one patient only- no standard deviation calculated | 0.25 (0.07)

4. Primary Outcome: Body Mass Index (BMI) in Control and Chronic Kidney Disease (CKD3b, CKD4, CKD5) Groups
Description: Body Mass Index (BMI) is calculated from subject's weight (kilogram) and height (meter)
Time Frame: This is a cross sectional study; only one measurement collected, termed "baseline"
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Control | Chronic Kidney Disease, Stage 5 (CKD5) | Chronic Kidney Disease, Stage 4 (CKD4) | Chronic Kidney Disease, Stage 3b (CKD3b)
Number analyzed (Participants) | 30 | 14 | 2 | 2
kg/m2 | 25.72 (4.42) | 29.51 (5.91) | 32.87 (6.01) | 26.83 (5.07)

5. Primary Outcome: Insulin Level in Control and Chronic Kidney Disease (CKD3b, CKD4, CKD5) Groups
Description: Insulin is a hormone made by the pancreas that allows the body to use or store sugar (glucose) from the food eaten. Insulin regulates blood sugar level.
Time Frame: This is a cross sectional study; only one measurement collected, termed "baseline"
Population: Data missing (1) for CKD4 and CKD5 group
Measure: Mean (Standard Deviation); unit: uU/mL
Arm/Group | Control | Chronic Kidney Disease, Stage 5 (CKD5) | Chronic Kidney Disease, Stage 4 (CKD4) | Chronic Kidney Disease, Stage 3b (CKD3b)
Number analyzed (Participants) | 30 | 13 | 1 | 2
uU/mL | 8.52 (5.74) | 8.02 (6.01) | 8.3 (NA) — only 1 patient, standard deviation is not calculated | 4.9 (1.56)

6. Primary Outcome: LCAT Activity (Lecithin-Cholesterol Acyltransferase) in Control and Chronic Kidney Disease Groups, Mainly to CKD3b, CKD4
Description: LCAT measures phospholipase activity in plasma. Measuring LCAT activity may be useful in clarifying the aspects of lipid metabolism in relation to reverse cholesterol transport
  No data collected- no standard deviation calculated
Time Frame: This is a cross sectional study; only one measurement collected, termed "baseline"
Population: Data not generated - due to insufficient number of patient recruited in CKD4 and CKD3b for comparison and analysis
Arm/Group | Control | Chronic Kidney Disease, Stage 5 (CKD5) | Chronic Kidney Disease, Stage 4 (CKD4) | Chronic Kidney Disease, Stage 3b (CKD3b)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Primary Outcome: CETP Activity (Lecithin-Cholesterol Acyltransferase) in Control and Chronic Kidney Disease Groups, Mainly to CKD3b, CKD4
Description: CETP activity measures the transfers of neutral lipids from high density lipoproteins (HDL) to very low density lipoprotein (VLDL) and low density lipoprotein (LDL). CETP may give us the other clue to lipoprotein metabolism and reverse cholesterol transport pathway
  No data collected- no standard deviation calculated
Time Frame: This is a cross sectional study; only one measurement collected, termed "baseline"
Population: Data not generated - due to insufficient number of patient recruited in CKD4 and CKD3b for comparison and analysis
Arm/Group | Control | Chronic Kidney Disease, Stage 5 (CKD5) | Chronic Kidney Disease, Stage 4 (CKD4) | Chronic Kidney Disease, Stage 3b (CKD3b)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: This is not an interventional study. No adverse event monitored.
Arm/Group | Control | Chronic Renal Disease (CKD3b) | Chronic Renal Disease (CKD4) | Chronic Renal Disease (CKD5)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination of study due to low number of enrollment in chronic kidney disease group 3b and 4.

Secondly, chronic kidney disease subjects prefer not to receive heparin. Heparin is necessary for our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2015-10-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT02755818/ICF_000.pdf
  • Study Protocol (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02755818/Prot_001.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT02755818/SAP_002.pdf